CLINICAL TRIAL: NCT02161861
Title: Improvement of IVF Fertilization Rates, by the Cyclic Tripeptide FEE - Prospective Randomized Study
Acronym: Fertiline
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the trial was discontinued for legislative reasons.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071002
Record Dates: First submitted 2014-04-28; First posted 2014-06-12 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Infertility; Pregnancy
Keywords: tripeptide FEE; fertilization rates; embryos; oocytes
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group cFEE (Experimental): The group cFEE will be similarly inseminated with 100000/ml motile spermatozoa and will be supplemented with cFEE 100µM during 18 hours.
  The cFEE will increase the fusiogenic capacities of a gamete,
  Interventions: Other: cFFE increase the fusiogenic capacities of a gamete
- untreated group (No Intervention): control group

INTERVENTIONS:
Other: cFFE increase the fusiogenic capacities of a gamete
  Other Names: The cyclic tripeptide
  Arms: group cFEE

SUMMARY:
cFEE peptide improves the IVF fertilization rate in mouse and fertilization index in human. It improves sperm movement's parameters.

It has been studied over 3 generations of mice and appears without any side effects. The Agence de la BioMédecine has given the authorization for testing the peptide in human IVF.

It is expected to improve the fertilization rate, and thus provide more embryos per IVF attempt.

160 couples will be included over 15 months. Patient sperm parameters should be suitable for IVF. Female should be between 18 and 43 year old. Each cohort of eggs will be randomly distributed to one of the 2 groups The first group will be inseminated with 100000/ml motile spermatozoa. The second will be similarly inseminated but in a middle which will be supplemented with cFEE 100µM.

Criteria: number of embryos in each group

DETAILED DESCRIPTION:
Name and address of the coordinating investigator : Prof. Jean Philippe Wolf, Histology - Embryology Department , Biology of Reproduction - . Cochin Hospital , 123 Bd Port Royal, 75014 Paris Promotor: AP- HP represented by DRCD - Hôpital Saint- Louis Inclusion Sites : CHU Cochin, Paris

Main objective:

- To improve fertilization rate in IVF by supplementation of culture media with a molecule increasing the sperm fertilizing ability.

Secondary objectives

* Compare the rates of cleavage between the two groups of zygotes
* Compare the percentage of good quality embryos

Number of patients : 160 Duration of the inclusion period : 15 months Duration of participation of the patient: For each couple, the duration of participation will be as many times nine months that pregnancies will be obtained from fresh or frozen embryo transfers.In the absence of pregnancy duration of participation will be only 15 days.

Time monitoring of children : 9 months

Total study duration : The total study duration will be 36 months

Rational :

The cyclic tripeptide FEEc reproduces the binding site of Fertilin Beta. It binds to the alpha 6 beta 1 integrin and increases sperm fertilizing ability, improving its movement's parameters . Added to insemination IVF media, it should increase fertilization rates .

Methodology:

Oocytes in each cohort will be divided into two groups, one of which will be inseminated with the control medium and the other group is inseminated in the presence of peptide. The fertilization rate and embryo quality will be compared between these two groups.

Statistical analysis:

In mice with healthy gamete, the observed fertilization rate increase in the presence of peptide was 100 %. The fertilization rate in human IVF is about 65%, male indications included. There is an improvement of the fertilization index of zona free human oocytes of about 90% . We can reasonably foresee an improvement of 15 % of the fertilization rate in normal IVF.

This is why we believe that the difference between fertilization rates of both treated and control groups must be meaningful for 160 attempts. In this calculation it was assumed that the intra cluster correlation (ie intra cohort oocyte ) resulted in a 'design effect' D equal to 4.

The analysis will include descriptive statistics for each quantitative parameter at each time : mean, standard deviation , minimum, maximum , median and quartiles , number of missing values . Quality parameters will be expressed by their frequency of distribution and associated 95% bilateral confidence intervals.The distributions of the numbers of blastomeres per embryo will be compared between the two groups by exact permutation test (stratified). This method is more suitable than "naive" comparison of these numbers, since it takes into account the possible correlation between results for embryos belonging to the same embryo cohort (Gibbons JD 1985 Non parametric statistical inference - Marcel Dekker New York ). The cellular index, the pregnancy rate, spontaneous abortions, therapeutic abortion, childbirth, will be compared using Student's t test and exact Fisher test. All tests will be bilateral, and look for possible negative effects, set at 5%. Calculations will be performed using SAS statistical software v9.13 (SAS Institute, Cary , NC) under the supervision of Professor Eric Vicaut URC Lariboisière St. Louis.

Primary endpoint : Rate of fertilization Expected Benefits : Improved fertilization rates of at least 15 %

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for in vitro fertilization except indication of ICSI. That is to say : the patients whose sperm has the following characteristics :

  * Sperm count over 107 spz /ml and Mobility * ( a + b ) is greater than 15 %
  * Typical forms above 10%
* Women aged 18 to 43 years.
* Patients gave their informed written consent
* People affiliated to a social security system

Exclusion Criteria:

* Patients whose sperm indicates the use or ICSI
* Patients who have not given their consent or without the consent of one of the two spouses
* Ovarian failure , menopause

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Fertilization rates | 24 hours

SECONDARY OUTCOMES:
Embryo quality | day 5
  The embryo quality will be assessed according to the number of blastomeres, the presence of cytoplasmic fragments, multinucleated blastomeres, they shape and regularity, and their cleavage rate. Data will be compared to the Z score classification for the zygote, and the Gardner classification for the blastocyste.
Pregnancy outcome | 9 months
Baby health | Year one
  Baby health will be assessed on data collected during the pregnancy by the OBGYN, the 6 month ultrasound examination, and the health of the baby at delivery. It will consider the APGAR index and its weight and stature. During the first year of life, the baby health will be assessed by the pediatrician's examination at 6 month and one year old.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-philippe Wolf, MD, Principal Investigator — Embryology Department , Biology of Reproduction - . Cochin Hospital
Locations (1):
- Wolf, Paris, France

REFERENCES:
- [Background] Yuan R, Primakoff P, Myles DG. A role for the disintegrin domain of cyritestin, a sperm surface protein belonging to the ADAM family, in mouse sperm-egg plasma membrane adhesion and fusion. J Cell Biol. 1997 Apr 7;137(1):105-12. doi: 10.1083/jcb.137.1.105. PMID 9105040
- [Background] Ziyyat A, Naud-Barriant N, Barraud-Lange V, Chevalier F, Kulski O, Lemkecher T, Bomsel M, Wolf JP. Cyclic FEE peptide increases human gamete fusion and potentiates its RGD-induced inhibition. Hum Reprod. 2005 Dec;20(12):3452-8. doi: 10.1093/humrep/dei241. Epub 2005 Aug 11. PMID 16096325
- [Background] Barraud-Lange V, Naud-Barriant N, Ducot B, Chambris S, Bomsel M, Wolf JP, Ziyyat A. Cyclic QDE peptide increases fertilization rates and provides healthy pups in mouse. Fertil Steril. 2009 May;91(5 Suppl):2110-5. doi: 10.1016/j.fertnstert.2008.05.088. Epub 2008 Aug 9. PMID 18692807
- [Background] Wolf JP, Bomsel M. Brevet international "Peptide augmentant la capacité fusiogène d'une gamète" Université Paris 13 et CNRS. N° d'enregistrement 03 13545 ; N° de publication 2 862 225. 2003